CLINICAL TRIAL: NCT02459600
Title: Methodes of Meausring Refraction in Children Under General Anesthesia
Brief Title: Comparison of Refraction Measurments in Children Under General Anesthesia, With and Without Cycloplegic Drops
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Zvi Gur MD, Zvi Gur, MD, Soroka University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SOR026014CTIL
Record Dates: First submitted 2015-05-05; First posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: General Anesthesia
Keywords: Eye surgery; Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All participants (Experimental): The measurement will be done at all the participants. the results will the divides in the following way:
  1. Refraction measurements under general anesthesia without cycloplegic eye drops.
  2. Refraction measurements under general anesthesia with cycloplegic eye drops.
  Interventions: Other: instulling cyclopentolate drops in the eye

INTERVENTIONS:
Other: instulling cyclopentolate drops in the eye — measuring refraction with and wirthout cyclopentolate drops under general anesthesia

SUMMARY:
Assessment of refraction measurements in children under general anesthesia, with or without cyclopelgic eye-drops

DETAILED DESCRIPTION:
Comparing to adults, children have high ability to preform accommodation of the intraocular lens, that is due to the Ciliary muscle. In order to measure children's refraction in an accurate way the Ciliary muscle must be paralyzed and that is usually done be cycloplegic eye-drops .In case a child is undergoing a medical procedure under general anesthesia the assumption that the Ciliary muscle is paralyzed (complete or partially) due to anesthetic medications. In this study we would like to compare the refraction measurements in children under who undergo general anesthesia before and after applying cycloplegic eye-drops. In this way we can learn about the effect of anesthetic medication on the Ciliary muscle.

ELIGIBILITY:
Inclusion Criteria:

1. 1 - 12 years old
2. Eyes that didn't underwent surgical procedure

Exclusion Criteria:

1. eye operation

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
difference in refraction results with and without cyclopentolate drops under general anesthesia | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Gur, MD, Principal Investigator — Soroka University Medial Center, Israel
Locations (1):
- Soroka, Beersheba, Israel